CLINICAL TRIAL: NCT03093857
Title: Investigation of the Cerebrospinal Fluid and Further Tissue Samples for Biomarker Indicating Spinal Ischemia and Organ Failure in Patients With Thoracoabdominal Aortic Aneurysm
Acronym: TAAA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-035
Record Dates: First submitted 2017-03-16; First posted 2017-03-28 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Determination of biomarker — Liquor, blood, and urine samples will be drawn and measured at different time points.

SUMMARY:
Patients with a thoracoabdominal aortic aneurysm in need of an endovascular or open operative restructuring will be asked to participate in this study. After obtaining written consent a central venous catheter and a liquor drainage will be routinely placed during surgery. The catheter and the drainage will stay in the patients for at least 72 hours postoperatively. In total, nine measurements of the liquor and serum will be performed within a week in order to determine the following parameters: neuropeptide P, neuropeptide Y, neurofilament triplet protein (NFL), S100B, glial fibrillary protein (GFAp), lactate, glucose, or oxygen.

DETAILED DESCRIPTION:
Patients with complex aortic diseases receiving an operative treatment are under risk of spinal cord damage due to insufficient blood circulation of the spinal cord during surgery. The risk depends on comorbidities, extent of surgery, and the perioperative management. Despite an adequate preoperative imaging, assessment of the blood circulation of the spinal cord during endovascular or open operative restructuring is struggling. Beside the monitoring possibilities of the spinal cord functions during surgery, insufficient approaches regarding early detection of spinal ischemia by using laboratory parameters exist. Several biomarker, e.g. neuropeptide P, neuropeptide Y, neurofilament triplet protein (NFL), S100B, glial fibrillary protein (GFAp), lactate, glucose, or oxygen, will be evaluated singularly or as a bundle of markers in small patient groups. Surgeries of thoracoabdominal aortic aneurysms are associated with high risks despite already existing high standardized procedures (Cowan et al. 2003). The major complications are cardiovascular, renal, pulmonary, gastrointestinal complications, and ischemias of the spinal cord. Especially, the ischemia of the spinal cord is a feared complication caused by the irreversibility and the small time frame.

During the study samples of liquor and tissues (serum, urine) will be drawn pre-, peri- and postoperatively. Patients will receive a routinely placed liquor drainage due to the temporal duration in surgery. The liquor drainage stays in the patient also in the early postoperative phase. Hence, the patient will not be bothered with additional examinations. Additionally, biomaterial (blood) will be drawn routinely and used for the biomarker measurement as well as biobanking.

ELIGIBILITY:
Inclusion Criteria:

* presence of thoracoabdominal aortic aneurysm
* endovascular or open operative restructuring
* age>18 years
* given written consent
* subjects, who are mentally and legally capable to understand the scope of the trial and comply with the protocol

Exclusion Criteria:

* local skin infection (cutaneous fungus, acne)
* pregnant or lactating females
* parallel participation in another clinical trial
* incarcerated subjects
* subjects, who are in an interdependency with the sponsor or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thoracoabdominal aortic aneurysm
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in neuropeptide P | baseline and postoperative day 1 and postoperative day 2 and week 1
Change in neuropeptide Y | baseline and postoperative day 1 and postoperative day 2 and week 1
Change in neurofilament triplet protein (NFL) | baseline and postoperative day 1 and postoperative day 2 and week 1
Change in S100B | baseline and postoperative day 1 and postoperative day 2 and week 1
Change in Glial fibrillary acidic protein (GFAp) | baseline and postoperative day 1 and postoperative day 2 and week 1
Change in lactate | baseline and postoperative day 1 and postoperative day 2 and week 1
Change in glucose | baseline and postoperative day 1 and postoperative day 2 and week 1
Change in oxygen | baseline and postoperative day 1 and postoperative day 2 and week 1

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Gombert, Dr. med., Principal Investigator — UK Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided